CLINICAL TRIAL: NCT06913296
Title: Do PTeye Score Correlate With Biochemical Markers in Parathyroid Adenoma?
Brief Title: PTeye in Parathyroid Adenoma
Status: Recruiting | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Papavramidis Theodossis, Professor of Surgery, Aristotle University Of Thessaloniki
Other Study IDs: PTeye adenoma
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Parathyroid Adenoma
Keywords: parathyroid adenoma; near-infrared autofluorescence
MeSH Terms: conditions — Parathyroid Neoplasms | interventions — Parathyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parathyroid adenoma patients: Patients undergoing surgery for parathyroid adenoma will be enrolled in this study. Parathyroid glands will be identified with the application of autofluorescence device PTeye and the values obtained by the device after parathyroid gland recognition will be registered.
  Interventions: Procedure: parathyroidectomy

INTERVENTIONS:
Procedure: parathyroidectomy — typical open parathyroidectomy

SUMMARY:
Identifying the parathyroids is compulsory for success of parathyroidectomy for parathyroid adenoma. Near-infrared autofluorescence devices have been proposed as useful intraoperative tools for the identification of parathyroid glands. The aim of the present study is to evaluate the correlation of PTeye autofluorescence device with biochemical data of parathyroid adenoma patients.

DETAILED DESCRIPTION:
Identifying the parathyroids is compulsory for success of parathyroidectomy for parathyroid adenoma. Near-infrared autofluorescence devices have been proposed as useful intraoperative tools for the identification of parathyroid glands. Two approaches are available to surgeons to perform near-infrared autofluorescence: (i) Camera-based systems (CBS) and (ii) Probe-based systems such as PTeye™ (Medtronic, Minneapolis, MN).The aim of the present study is to evaluate the correlation of PTeye autofluorescence device with biochemical data of parathyroid adenoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* primary hyperparathyroidism caused by adenoma
* patient's informed consent acquired

Exclusion Criteria:

* Secondary and tertiary hyperparathyroidism
* Re-operation for adenoma
* Previous neck surgery
* Patient enrolled in another study that may affect the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for parathyroid adenoma
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
assess the correlation of PTeye values with biochemical data | intraoperatively and 1st postoperative day
  Biochemical data included are pre- and postoperative parathyroid hormone, serum calcium, phosphorus and vitamin D levels

CONTACTS AND LOCATIONS:
Overall Officials: Moysis Moysidis, Dr, Study Chair — Euromedica Kyanos Stavros; Chrysa Papadopoulou, Study Chair — Euromedica Kyanos Stavros
Locations (1):
- Aristotle Univeristy of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No